CLINICAL TRIAL: NCT02251912
Title: Oxytocin Treatment of Alcohol Dependence: A Randomized, Placebo-Controlled Trial
Brief Title: Oxytocin Treatment of Alcohol Dependence
Acronym: OTETOH-3
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 12-1862b; 1R21AA021927-01A1 (NIH)
Record Dates: First submitted 2014-09-25; First posted 2014-09-29 (Estimated); Results first posted 2017-08-15 (Actual); Last update posted 2017-08-15 (Actual); Status verified 2017-05

CONDITIONS: Alcohol Dependence
Keywords: Alcohol dependence; Alcohol; Oxytocin; Intranasal administration
MeSH Terms: conditions — Alcoholism

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active (Experimental): Intranasal oxytocin doses 2-3 times/day for 12 weeks
  Interventions: Drug: Intranasal Oxytocin
- Control (Placebo Comparator): Intranasal placebo doses 2-3 times/day for 12 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Intranasal Oxytocin — 10 insufflations (40IU of oxytocin total) given 3 initially then 2 times daily for 12 weeks
  Other Names: Syntocinon spray
  Arms: Active
Drug: Placebo — 10 insufflations (same solution as active treatment minus oxytocin) given 3 initially and then 2 times daily for 12 weeks
  Arms: Control

SUMMARY:
Purpose: Test whether oxytocin treatment decreases drinking in people who have been consuming alcohol heavily for long periods and are physically and psychologically dependent on alcohol.

Participants: 50 adults with alcohol dependence

Procedures (methods): Oxytocin or placebo will be administered three times a day for the first 2 days followed by twice daily intranasal doses for the rest of the 12 weeks. Before, during and at the end of the trial, each subject will undergo evaluations including breathalyzer readings, rating withdrawal symptoms, interviews about amount of alcohol consumed since last clinic visit, subject self-ratings of anxiety, alcohol craving and, at some visits, laboratory measures (blood and urine) to monitor safety and alcohol/drug use. Following the active phase of the trial, subjects will be followed up at 4 weeks and 12 weeks to evaluate for post-medication safety and efficacy

DETAILED DESCRIPTION:
The purpose of this research study is to learn whether oxytocin treatment decreases drinking and alcohol craving in people who have been consuming alcohol heavily for long periods and are unable to stop drinking on their own. Oxytocin is made naturally and is released in parts of the brain where it acts like a chemical signal from one cell to another. Oxytocin is approved by the Food and Drug Administration for stimulating labor in pregnant women but is not approved as a treatment to decrease alcohol drinking.

People who drink large amounts of alcohol every day or many days per week for weeks or months undergo chemical changes in their brains. They continue to drink frequently and heavily because, even though they may know drinking is not good for their health, they experience unpleasant symptoms if they stop or decrease drinking. Those symptoms can include increased anxiety, difficulty sleeping, difficulty tolerating stress, mild to moderate withdrawal symptoms such as tremors, nausea, feeling sweaty and/or headaches, and cravings to drink. Studies found that giving oxytocin to alcohol-addicted animals reduced symptoms when they were put into alcohol withdrawal. A pilot study conducted at UNC found that twice daily intranasal doses of oxytocin decreased withdrawal symptoms in heavy drinkers who were admitted to a hospital for medical detoxification to come off alcohol.

This study will test whether daily intranasal oxytocin treatment for 12 weeks will decrease how much subjects drink as well as craving for alcohol and anxiety.

Prospective subjects must have been drinking large amounts of alcohol for a sustained period to qualify for this study and want help to stop or cut back on their drinking. Subjects will self-administer oxytocin or placebo in this study in an intranasal spray. The placebo spray contains all of the ingredients of the oxytocin spray EXCEPT oxytocin. Subjects' assignment to oxytocin or placebo treatment will be random (like a flip of a coin).

Subjects must sign a consent form to take part in this study. Their participation in the study will last up to 14-15 weeks. Prospective subjects will be recruited from the community through advertisements (radio, social media, mass emails, etc). Those who respond to advertisements will undergo initial screening over the phone. Prospective subjects who appear to meet study criteria based on the phone screen will give informed consent and undergo more detailed evaluation during a screening clinic visit. If they are found to meet study criteria, they will shortly thereafter attend another clinic visit (randomization clinic visit) during which they will be randomized to oxytocin or placebo treatment and take their first test dose under study personnel supervision. They will then take home the bottle contained the intranasal study medication to which they have been randomized and self-administer intranasal test doses at home for the remainder of the 12-week test treatment period. New intranasal spray bottles will be exchanged for old every 2 weeks. Subjects will attend 8 additional clinic visits over a 12 week period after the randomization clinic visit. Each clinic visit will last 1-2 hours.

Procedures during screening clinic visits will include: 1) a Breathalyzer test (a reading of zero is necessary for subjects to give informed consent); 2) vital sign measures and a CIWA (Clinical Institute Withdrawal Assessment for Alcohol) scale score (subjects must not be in significant withdrawal when they give informed consent and undergo screening evaluations); 3) urine collection to test for addictive substances and pregnancy; 4) completion of the Time Line Follow Back (TLFB) interview to determine how many standard drinks have been consumed during the previous 90 days; 5) interview using the Structured Clinical Interview for DSM-IV (SCID). Alcohol use module to confirm subjects meet DSM-IV TR criteria for alcohol dependence; 6) completion of the MINI International Neuropsychiatic Interview (MINI) diagnostic sections on substance use disorders, psychotic disorders, bipolar disorder, and eating disorders; 7) subject completion of the Penn Alcohol Craving Scale (PACS); 8) subject completion of the Spielberger State-Trait Anxiety Inventory (SSTAI); 9) physical examination by a study doctor; 10) blood collection for laboratory tests.

During the randomization clinic visit, subjects who screen into the study will be randomly assigned (like the flip of a coin) to receive either oxytocin or placebo intranasal spray. Members of the researcher staff will instruct subjects in how to self-administer intranasal spray doses from a spray bottle. Subjects will then take their first intranasal test dose during a clinic visit scheduled shortly after this screening visit. Subjects will take an intranasal spray bottle home with them after this visit and continue to self-administer intranasal test doses three time each day (at approximately breakfast, lunch and dinner time) for two days and thereafter will take intranasal test doses twice each day (at approximately breakfast and dinner time). Each dose will be 10 sprays into their nose (5 per nostril alternating between nostrils).

Procedures during subsequent outpatient clinic visits will include: 1) a Breathalyzer reading; 2) vital signs and a CIWA score; 3) a TLFB interview; 4) PACS self-rating; 5) State portion of the SSTAI (SSAI) self-rating; 6) at the week 4, 8, and 12 clinic visits, blood and urine collection for laboratory tests, pregnancy tests and addictive drug screens.

During the randomization clinic visit and each subsequent clinic visit, subjects' Breathalyzer reading must be less than .04 g/dL for study procedures to be done. If Breathalyzer readings are higher, the visit will be rescheduled. Also, during each of these clinic visits, a Medical Management session (special talk therapy for alcohol dependence) will be conducted with the study doctor before patients are discharged.

ELIGIBILITY:
Inclusion Criteria:

* Meeting criteria for DSM-IV-TR alcohol dependence.
* Consumption of at least 35 standard drinks/week for men or 28 standard drinks/week for women for at least 4 consecutive weeks prior to enrollment into the study.
* Women who are able to conceive children and who are sexually active must be on an effective form of birth control such as oral contraceptives, IUDs or the use of condoms with spermicide.
* Competency to give valid informed consent as indicated by a) a Breathalyzer reading at the time the consent form is signed showing an estimated blood alcohol level (BAL) of zero; b) ability to understand the written informed consent form demonstrated by correctly answering questions about the contents of the form after reading the consent form without help (this will also determine whether prospective subjects can read and understand the study questionnaires).
* Ability to get to appointments either through personal or public transportation.
* Ages 18-65.

Exclusion Criteria:

* History of alcohol withdrawal-related seizures, delirium tremens or hallucinations.
* Clinically significant medical disease that might interfere with the evaluation of the study medication or present a safety concern (e.g., renal insufficiency, cirrhosis, unstable hypertension, unstable diabetes mellitus, seizure disorder).
* History of psychotic disorder or admission for mania, meeting criteria for an eating disorder in the last 2 years, current moderate or severe major depression, current suicidal ideation.
* Currently meeting DSM-IV TR criteria for dependence on addictive substances other than alcohol except for nicotine or caffeine. Substance abuse disorders are not exclusionary.
* Consumption during the week prior to enrollment or plans to consume during the 12-week trial of benzodiazepines, barbiturates, anticonvulsants or stimulants.
* AST or ALT > 5 times ULN, bilirubin > 1.5 X ULN, sodium < 132 or > 150 mMol/L, potassium < 3.2 or > 5.3 mMol/L.
* Women who are pregnant or breastfeeding.
* Currently participating in or intent to participate in an additional alcohol treatment program during the study period other than Alcoholics Anonymous.
* Court-mandated participation in alcohol treatment or pending incarceration.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2015-07 (Actual); Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cort A Pedersen, MD, Principal Investigator — University of North Carolina, Chapel Hill; James C Garbutt, MD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Active | Control
Started | 12 | 10
Completed | 10 | 5
Not Completed | 2 | 5
Not completed — Withdrawal by Subject | 2 | 3
Not completed — Adverse Event | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Active | Control | Total
Number analyzed (Participants) | 12 | 10 | 22
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 12 | 10 | 22
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 4 | 9
  Male | 7 | 6 | 13
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 2 | 3
  White | 11 | 8 | 19
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 12 | 10 | 22

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Heavy Drinking Days
Description: Mean proportion of days per week, over the 12-week trial, when subjects drank heavily (5 or more standard drinks for men, 4 or more standard drinks for women).
Time Frame: 12 weeks
Measure: Least Squares Mean (Standard Error); unit: proportion of days per week
Arm/Group | Active | Control
Number analyzed (Participants) | 12 | 10
proportion of days per week | 0.3072 (0.094) | 0.5914 (0.1024)

2. Primary Outcome: Mean Weekly Drinks Per Drinking Day
Description: The mean number of standard drinks (the amount of alcohol in a standard drink is roughly equivalent to the amount of alcohol in a 12 ounce beer) consumed by subjects on days when they drank alcoholic beverages each week averaged over the 12-week trial.
Time Frame: 12 weeks
Measure: Least Squares Mean (Standard Error); unit: number of drinks per drinking day
Arm/Group | Active | Control
Number analyzed (Participants) | 12 | 10
number of drinks per drinking day | 4.8929 (0.5868) | 7.5621 (0.6108)

3. Secondary Outcome: Alcohol Craving
Description: Mean weekly Penn Alcohol Craving Scale (PACS) scores.The PACS is a five-item self-administered instrument for assessing craving, frequency, intensity, and duration of thoughts about drinking as well as the ability to resist drinking. Scores range from: Minimum: 0 Maximum: 30 Lower scores are associated with better outcomes.
Time Frame: 12 weeks
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Active | Control
Number analyzed (Participants) | 12 | 10
units on a scale | 10.8481 (2.1254) | 12.6685 (2.3122)

ADVERSE EVENTS:
Arm/Group | Active | Control
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/10
Other Adverse Events (participants affected / at risk) | 0/12 | 2/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active (N=12) | Control (N=10)
sore throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) — backflow of intranasal spray down the throat was reported to cause soreness in the pharyngeal area
nosebleed (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) — a nosebleed associated with repeated intranasal administration of test substance that did not recur after subject stopped intranasal doses

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No